CLINICAL TRIAL: NCT04008797
Title: An Open-label Study of E7386 in Combination With Other Anticancer Drug(s) in Subjects With Solid Tumors
Brief Title: A Study of E7386 in Combination With Other Anticancer Drug(s) in Participants With Solid Tumor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E7386-J081-102; 2022-003300-32 (EudraCT Number); 2023-510275-64-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2019-06-24; First posted 2019-07-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Neoplasms; Neoplasms; Carcinoma, Hepatocellular; Liver Neoplasms; Colorectal Neoplasms
Keywords: Endometrial cancer; Solid Tumor; Hepatocellular carcinoma; Colorectal cancer; E7386; Lenvatinib
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms; Carcinoma, Hepatocellular; Liver Neoplasms; Colorectal Neoplasms | interventions — E-7386; lenvatinib; Doxorubicin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: The Dose Optimization part and HCC subpart of Expansion part of the study are randomized. The Dose Escalation part, and CRC/EC subparts of Dose Escalation part are non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Dose Escalation Part: HCC: E7386 QD Subpart + Lenvatinib (Experimental): Participants with hepatocellular carcinoma (HCC) will receive E7386, once daily (QD) for 5 or 6 consecutive days followed by a period of time without treatment in Cycle 0 (6 or 7 days). Participants with HCC will receive E7386, QD in combination with lenvatinib 8 milligram (mg) (participants with body weight of less than [<] 60 kilograms [kg]) or 12 mg (participants with body weight >=60 kg), capsules, orally, QD in 28-day treatment cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386; Drug: Lenvatinib
- Dose Escalation Part: HCC: E7386 BID Subpart + Lenvatinib (Experimental): Participants with HCC will receive E7386, twice daily (BID) for 5 or 6 consecutive days in Cycle 0 (6 or 7 days). Participants with HCC will receive E7386, BID in combination with lenvatinib 8 mg (participants with body weight of < 60 kg) or 12 mg (participants with body weight >=60 kg) capsules, orally, QD in 28-day treatment cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386; Drug: Lenvatinib
- Dose Escalation Part: Other ST: E7386 QD Subpart + Lenvatinib (Experimental): Participants with solid tumor (ST) (except for HCC) will receive E7386, QD for 5 or 6 consecutive days followed by a period of time without treatment in Cycle 0 (6 or 7 days). Participants with ST (except for HCC) will receive E7386, QD in combination with lenvatinib 20 mg, capsules, orally, QD in 28-day treatment cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386; Drug: Lenvatinib
- Dose Escalation Part: Other ST: E7386 BID Subpart + Lenvatinib (Experimental): Participants with ST (except for HCC) will receive E7386, BID for 5 or 6 consecutive days in Cycle 0 (6 or 7 days). Participants with ST (except for HCC) will receive E7386, BID in combination with lenvatinib 20 mg, capsules, orally, QD in 28-day treatment cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386; Drug: Lenvatinib
- Dose Expansion Part: HCC Subpart: Lenvatinib Only (Experimental): Participants with HCC will receive lenvatinib 8 mg (participants with body weight of <60 kg) or 12 mg (participants with body weight >=60 kg), capsules, orally, QD in 28-day treatment cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program
  Interventions: Drug: Lenvatinib
- Dose Expansion Part: HCC Subpart: E7386 + Lenvatinib (Experimental): Participants with HCC will receive lenvatinib 8 mg (participants with body weight of <60 kg) or 12 mg (participants with body weight >=60 kg), capsule, orally QD in combination with E7386 y, BID in 28-day treatment cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386; Drug: Lenvatinib
- Dose Expansion Part: CRC Subpart: E7386 + Lenvatinib (Experimental): Participants with colorectal cancer (CRC) will receive E7386, BID in combination with lenvatinib 20 mg, capsules, orally, QD in 28-day treatment cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386; Drug: Lenvatinib
- Dose Expansion Part: EC Subpart: E7386 + Lenvatinib (Experimental): Participants with endometrial cancer (EC) will receive E7386, BID in combination with lenvatinib 14 mg, capsules, orally, QD in 28-day treatment cycles until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386; Drug: Lenvatinib
- Dose Optimization Part: EC Participants (Experimental): Participants with EC will be randomized to receive 2 different doses of E7386 in combination with lenvatinib capsule or lenvatinib capsule monotherapy in 28-days cycles, or treatment of physician's choice (TPC; doxorubicin in 21-day cycles or paclitaxel in 28-day cycles [3 weeks on/1 week off]), until PD, development of unacceptable toxicity, participant request to discontinue, withdrawal of consent, or termination of the study program.
  Interventions: Drug: E7386; Drug: Lenvatinib; Drug: Doxorubicin; Drug: Paclitaxel

INTERVENTIONS:
Drug: E7386 — E7386 dosing.
  Arms: Dose Escalation Part: HCC: E7386 BID Subpart + Lenvatinib; Dose Escalation Part: HCC: E7386 QD Subpart + Lenvatinib; Dose Escalation Part: Other ST: E7386 BID Subpart + Lenvatinib; Dose Escalation Part: Other ST: E7386 QD Subpart + Lenvatinib; Dose Expansion Part: CRC Subpart: E7386 + Lenvatinib; Dose Expansion Part: EC Subpart: E7386 + Lenvatinib; Dose Expansion Part: HCC Subpart: E7386 + Lenvatinib; Dose Optimization Part: EC Participants
Drug: Lenvatinib — Lenvatinib dosing.
  Other Names: Lenvima; E7080
Drug: Doxorubicin — Doxorubicin dosing.
  Arms: Dose Optimization Part: EC Participants
Drug: Paclitaxel — Paclitaxel dosing.
  Arms: Dose Optimization Part: EC Participants

SUMMARY:
The primary objective of this study is to assess the safety and tolerability and to determine the recommended Phase 2 dose (RP2D) of E7386 in combination with other anticancer drug(s), and to determine the optimal dose of E7386 in combination with lenvatinib in endometrial carcinoma (EC) (for EC Dose Optimization Part only).

DETAILED DESCRIPTION:
The Dose Escalation and Dose Expansion parts of the study have completed enrollment. The Dose Optimization part of the study is enrolling participants with endometrial carcinoma (EC) only.

ELIGIBILITY:
Inclusion Criteria:

1. HCC part only:

   Participants with confirmed diagnosis of unresectable HCC with any of the following criteria:
   1. Histologically or cytologically confirmed diagnosis of HCC, excluding fibrolamellar, sarcomatoid or mixed cholangio-HCC tumors
   2. Clinically confirmed diagnosis of HCC according to American Association for the Study of Liver Diseases (AASLD) criteria, including cirrhosis of any etiology and/or chronic hepatitis B or C infection

   ST part only (except for HCC):

   Participants with histologically or cytologically confirmed diagnosis of solid tumor for which no alternative standard therapy or no effective therapy exists
2. Life expectancy of >=12 weeks
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
4. All AEs due to previous anti-cancer therapy have either returned to Grade 0 to 1 except for alopecia or up to Grade 2 peripheral neuropathy (renal/bone marrow/liver function should meet the inclusion criteria)
5. Adequate washout period before study drug administration:

   1. Chemotherapy and radiotherapy: 3 weeks or 5 times the half-life, whichever is shorter
   2. Any antitumor therapy with antibody: 4 weeks or more
   3. Any investigational drug or device: 4 weeks or more
   4. Blood/platelet transfusion or granulocyte colony-stimulating factor (G-CSF): 2 weeks or more Note: Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not had radiation pneumonitis
6. Adequate controlled blood pressure (BP), renal function, bone marrow function, liver function, and serum mineral level
7. At least one measurable lesion based on mRECIST (for HCC Subparts in Dose Escalation Part) or on RECIST 1.1 (for Other ST Subparts in Dose Escalation Part and all subparts in Expansion and Dose Optimization Parts) meeting following criteria

   * At least 1 lesion of >=1.0 centimeter (cm) in the longest diameter for a non-lymph node or >=1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to RECIST 1.1 using computerized tomography (CT)/magnetic resonance imaging (MRI)
   * Lesions that have had external beam radiotherapy or loco-regional therapies such as radiofrequency ablation, or transarterial chemoembolisation (TACE)/ transarterial embolization (TAE) must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion
8. For HCC participants only: Child-Pugh score A. Note: If Child-Pugh score 7 or more was observed during Screening or Baseline, the participant is ineligible and re-assessment of the Child-Pugh score is not permitted
9. For HCC participants only: Participants categorized to stage B (not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment), or stage C based on Barcelona Clinic Liver Cancer (BCLC) staging system
10. For HCC Subpart in Expansion Part only: prior systemic therapy for locally advanced or metastatic disease is as defined below

    a. Participants who have received only one prior line of immuno oncology (IO) based regimen and have progressed on or after prior treatment with IO based regimen, or IO ineligible participants who have received no prior systemic therapy. Participants who previously received lenvatinib treatment are ineligible
11. For CRC Subpart in Expansion Part only: participants must have received at least 2 prior regimens (not exceeding 4 prior regimens) or could not tolerate standard treatment and must have received the following prior therapies in the metastatic setting if approved and locally available (progressed on at least 1 prior regimen in the metastatic setting or could not tolerate standard treatment):

    Note: Adjuvant chemotherapy counts as prior systemic treatment if there is documented disease progression within 6 months of treatment completion Note: If a participant is determined to be intolerant to prior standard treatment, the participant must have received at least of 2 cycles of that therapy Note: Participants who have received oral tyrosine kinase inhibitor (example, regorafenib) are ineligible
    1. Fluoropyrimidine, irinotecan and oxaliplatin with or without an anti-Vascular endothelial growth factor (VEGF) monoclonal antibody (mAb) (example, bevacizumab) Note: Capecitabine is acceptable as equivalent to fluoropyrimidine in prior treatment Note: Participants who have previously received fluoropyrimidine, oxaliplatin, and irinotecan as part of the same and only chemotherapy regimen, example, FOLFOXIRI or FOLFIRINOX, may be eligible after discussion with the Sponsor
    2. Chemotherapy with anti- epidermal growth factor receptor (EGFR) mAb (cetuximab or panitumumab) for participants with rat sarcoma virus (RAS) (Kirsten rat sarcoma viral oncogene homolog [KRAS)/ NRAS]) wild type (WT) CRC Note: RAS (KRAS/NRAS) WT participants with right or left CRC lesions who may have not been treated with anti-EGFR mAb based on local guidelines are eligible
    3. BRAF inhibitor (in combination with cetuximab ± binimetinib) for BRAF V600E mutated tumors
    4. Immune checkpoint inhibitor for participants with microsatellite instability-high (MSI-H) CRC
12. For EC Subpart in Expansion Part only: Participants must have EC that has progressed after prior platinum-based chemotherapy and an anti-programmed cell death (ligand) 1 (PD-[L])1)-directed therapy for EC (participants ineligible for IO therapy who have progressed after prior platinum-based chemotherapy are eligible). Up to 3 prior systemic therapies, of which up to 2 for metastatic or locally advanced disease, are permitted Note: There is no restriction regarding prior hormonal therapies For Dose Optimization Part only: Participants must have EC that has progressed after prior platinum-based chemotherapy and an anti-PD-(L)1-directed therapy for EC. Up to 3 lines of prior therapy, regardless of setting, are allowed. Participants must be eligible for treatment with either single-agent paclitaxel or single-agent doxorubicin as determined by the investigator, with consideration of previous therapies received for EC. Note: Prior hormonal therapy and radiation are allowed and do not count as prior lines of therapy.

Exclusion Criteria:

1. Any of cardiac conditions as follows:

   * Heart failure New York Heart Association (NYHA) Class II or above
   * Prolongation of QT interval with Fridericias correction (QTcF) to greater than (>) 480 millisecond (msec)
   * Left ventricular ejection fraction (LVEF) less than (<) 50 percent (%)
2. Major surgery within 21 days or minor surgery (that is, simple excision) within 7 days prior to starting study drug. Participant must have recovered from the surgery related toxicities to less than Grade 2 Note: Adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility
3. Known to be human immunodeficiency virus (HIV) positive Note: the sponsor has evaluated whether to include participant with HIV. Given that this is the first combination study of E7386 with lenvatinib and that the main mechanism of action of E7386 is immunomodulation of the tumor microenvironment along with the fact that several anti-retroviral therapies have drug-drug interaction with cytochrome P450 3A (CYP3A) substrates, the sponsor has decided not to include these participants at the current time. However, further considerations will be made moving forward based on new emerging data Note: HIV testing is required at screening only when mandated by local health authority
4. Participants with proteinuria on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein >=1 gram per 24 hour will be ineligible
5. Active infection requiring systemic treatment (Except for Hepatitis B and/or C [HBV/HCV] infection in HCC participants)

   In case of HBsAg (+) participants in HCC participants:
   * Antiviral therapy for HBV is not ongoing
   * HBV viral load is 2000 international unit per milliliter (IU/mL) or more at the Screening Period although antiviral therapy for HBV is ongoing
   * Has dual active HBV infection (HBsAg (+) and/or detectable HBV deoxyribonucleic acid [DNA]) and HCV infection (anti-HCV Ab (+) and detectable HCV ribonucleic acid [RNA]) at study entry
6. Diagnosed with meningeal carcinomatosis
7. Participants with central nervous system metastases are only eligible if they have been previously treated and are radiologically stable, (that is, without evidence of progression for at least 4 weeks prior to first dose of study treatment by repeat imaging), clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment
8. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen
9. Any of bone disease/conditions as follows:

   * T-score of < minus (-) 3.0 at the left or right total hip, left or right femoral neck or lumbar spine (L1-L4) as determined by dual energy x-ray absorptiometry (DXA) scan. Participants with T-score <-2.5 to -3.0 can only be included if treatment with a bisphosphonate (example, zoledronic acid) or denosumab has been started at least 14 days and no more than 6 months prior to the first dose of study drug
   * Metabolic bone disease, such as hyperparathyroidism, Paget's disease or osteomalacia
   * Symptomatic hypercalcemia requiring bisphosphonate therapy
   * History of any fracture within 6 months prior to starting study drug
   * Bone metastasis requiring orthopedic intervention
   * Bone metastasis not being treated by bisphosphonate or denosumab. Participants may be included if treatment with bisphosphonate or denosumab has been started at least 14 days prior to the first dose of study drug. Participants with previous solitary bone lesions controlled with radiotherapy are eligible
   * History of symptomatic vertebral fragility fracture or any fragility fracture of the hip, pelvis, wrist or other location (defined as any fracture without a history of trauma or because of a fall from standing height or less)
   * Moderate (25% to 40% decrease in the height of any vertebrae) or severe (>40% decrease in the height of any vertebrae) morphometric vertebral fracture at baseline
10. History of malignancy (except for original disease, or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, carcinoma in-situ [example, bladder or cervix]) within the past 24 months prior to the first dose of study drug
11. For HCC Subpart in Dose Escalation Part only: Participants who experienced discontinuation of lenvatinib, 2 or more dose reductions of lenvatinib required from initial dose level of this study due to its toxicity, or participants who experienced single dose reduction or consecutive >=8 days dose interruption of lenvatinib within 60 days from the first dose, due to its toxicity. HCC Subpart in Expansion Part only: Participants who previously received lenvatinib treatment are ineligible.

    EC Subpart in Expansion Part only: Participants previously treated with lenvatinib who experienced discontinuation of lenvatinib due to toxicity, or dose reduction to less than 10 mg of lenvatinib due to toxicity within 60 days from the first dose.

    EC Dose Optimization Part only: Participants who previously received lenvatinib treatment are ineligible.
12. Bleeding or thrombotic disorders or use of anticoagulants requiring therapeutic International Normalized Ratio (INR) monitoring for HCC participants only (example, warfarin or similar agents). Treatment with low molecular weight heparin and factor X inhibitors is permitted. Treatment with antiplatelet agents is prohibited for HCC participants in Dose Escalation Part only
13. Gastrointestinal bleeding event or active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug
14. For HCC participants only: History of hepatic encephalopathy within 6 months prior to starting study drug
15. For EC Subpart in Expansion and Dose Optimization Parts only: carcinosarcoma (malignant mixed Mullerian tumor), endometrial leiomyosarcoma, and endometrial stromal sarcomas
16. Has preexisting >=Grade 3 gastrointestinal or non-gastrointestinal fistula
17. Evidence of current Coronavirus disease 2019 (COVID-19) infection or ongoing unrecovered active sequelae of COVID-19 infection
18. Males who have not had a successful vasectomy (confirmed azoospermia) if their female partners meet the exclusion criteria above (that is, the female partners are of childbearing potential and are not willing to use a highly effective contraceptive method throughout the study period and after study drug discontinuation). No sperm donation is allowed during the study period and after study drug discontinuation
19. Has a known psychiatric or substance abuse disorder that would interfere with the participant ability to cooperate with the requirements of the study
20. Evidence of clinically significant disease (example, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator could affect the participant safety or interfere with the study assessments
21. Scheduled for major surgery during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Part: Number of Participants with Dose-limiting Toxicities (DLTs) | Cycle 0 (Cycle 0 length=6 or 7 days) up to Cycle 1 (Cycle 1 length=28 days)
  DLTs will be defined as any of the events that are considered by the investigator to be at least possibly related to therapy with the study medication. Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE 5.0).
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 30 days after the last dose of study drug or before initiating post anti-cancer treatment (up to approximately 90 months)
Dose Optimization Part: Objective Response Rate (ORR) per RECIST 1.1 by Investigator Assessment | From first dose of study drug until PD, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 90 months)
  The ORR is defined as the percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR). The ORR will be assessed by investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for dose optimization part.

SECONDARY OUTCOMES:
Dose Escalation Part: Cmax: Maximum Observed Plasma Concentration for E7386 | Day 1 to Day 8
Dose Escalation Part: Cmax: Maximum Observed Plasma Concentration for Lenvatinib | Day 8
Dose Escalation Part: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for E7386 | Day 1 to Day 8
Dose Escalation Part: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Lenvatinib | Day 8
Dose Escalation Part: AUC: Area Under the Plasma Concentration Versus Time Curve for E7386 | Day 1 to Day 8
Dose Escalation Part: AUC: Area Under the Plasma Concentration Versus Time Curve for Lenvatinib | Day 8
Dose Escalation Part: CL/F: Apparent Total Body Clearance for E7386 | Day 1 to Day 8
Dose Escalation Part: CL/F: Apparent Total Body Clearance for Lenvatinib | Day 8
Dose Escalation Part: Vz/F: Apparent Volume of Distribution for E7386 | Day 1 to Day 8
Dose Escalation Part: Vz/F: Apparent Volume of Distribution for Lenvatinib | Day 8
Percentage of Participants with Best Overall Response (BOR) | From first dose of study drug until progression of disease (PD), development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 90 months)
  BOR is defined as confirmed CR, confirmed PR, stable disease (SD), PD, and not evaluable (NE). The BOR will be assessed by investigator based on Modified Response Evaluation Criteria in Solid Tumors (mRECIST) for HCC subparts in dose escalation part and based on RECIST version 1.1 for ST subparts in dose escalation part, and for HCC subpart, CRC subpart, EC subpart in dose expansion part and in dose optimization part.
Objective Response Rate (ORR) | From first dose of study drug until PD, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 90 months)
  The ORR is defined as the percentage of participants with a BOR of CR or PR. The ORR will be assessed by investigator based on mRECIST for HCC subparts in dose escalation part and based on RECIST version 1.1 for ST-subparts in dose escalation part, and for HCC subpart, CRC subpart, EC subpart in dose expansion part.
Disease Control Rate (DCR) | From first dose of study drug until PD, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 90 months)
  DCR is defined as the percentage of participants with a BOR of CR, PR, or SD. The DCR will be assessed by investigator based on mRECIST for HCC subparts in dose escalation part and based on RECIST version 1.1 for ST-subparts in dose escalation part, and for HCC subpart, CRC subpart, EC subpart in dose expansion part and in dose optimization part.
Clinical Benefit Rate (CBR) | From first dose of study drug until PD, development of unacceptable toxicity, participant requests to discontinue, withdrawal of consent or study termination (up to approximately 90 months)
  The CBR is defined as the percentage of participants with a BOR of CR, PR, or durable SD. The CBR will be assessed by investigator based on mRECIST for HCC subparts in dose escalation part and based on RECIST version 1.1 for ST-subparts in dose escalation part, and for HCC subpart, CRC subpart, EC subpart in dose expansion part and in dose optimization part.
Progression-free Survival (PFS) | From first dose of study drug until PD, or death from any cause, whichever occurs first (up to approximately 90 months)
  PFS is defined as the time from the date of the first dose to the date of the first documentation of confirmed PD or death, whichever occurs first. The PFS will be assessed by investigator based on mRECIST for HCC subparts in dose escalation part and based on RECIST version 1.1 for ST-subparts in dose escalation part, and for HCC subpart, CRC subpart, EC subpart in dose expansion part and in dose optimization part.
Overall Survival (OS) | From first dose of study drug until death from any cause (up to approximately 90 months)
  OS is defined as the time from the first dose of study drug to death due to any cause. OS will be calculated for all subparts in dose expansion part, dose optimization part, and HCC subparts in dose escalation part only.
Duration of Response (DOR) | From first dose of study drug until PD, or death from any cause, whichever occurs first (up to approximately 90 months)
  DOR is defined as the time from the first documentation of PR or CR to the first documentation of disease progression or death due to any cause (whichever occurs first). DOR will be calculated for all subparts in dose expansion part, dose optimization part, and HCC subparts in dose escalation part only.

CONTACTS AND LOCATIONS:
Locations (107):
- United States (28):
  - UAMS, Little Rock, Arkansas
  - University of California San Diego (UCSD) - Moores Cancer Center(All), La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Pasadena Liver Center, Pasadena, California
  - California Pacific Medical Center, San Francisco, California
  - UCLA University of California - Los Angeles, Santa Monica, California
  - John Muir Clinical Research, Walnut Creek, California
  - University of Colorado Cancer Center - Anschutz Medical Campus, Aurora, Colorado
  - Uni. Of Miami- Sylvester Cancer Centre, Miami, Florida
  - Florida Cancer Specialists - South, Sarasota, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Women's Cancer Care - Covington, LA, Covington, Louisiana
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Perlmutter Cancer Center- NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center (MMC) - Jack D. Weiler Hospital, The Bronx, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Centre, Sioux Falls, South Dakota
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center (VUMC) - Vanderbilt-Ingram Cancer Center (VICC) - Nashville, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas Southwestern Medical, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson/University of Washington Cancer Consortium, Seattle, Washington
- Canada (3):
  - Sunnybrook Research Institute, Toronto, Ontario
  - CHUM, Unit for Innovative Therapies, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- China (13):
  - Beijing Cancer Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Sun Yan-sen University Cancer Center, Guangzhou
  - Sun Yat-Sen Memrial Hospital, Sun Yat-Sen University, Guangzhou
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Fudan University Cancer Center, Shanghai
  - The Tenth People's Hospital; Shanghai Tongji University, Shanghai
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
  - Tianjin Cancer Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
- Odense University Hospital, Odense, Denmark
- France (23):
  - CHU Amiens-Picardie (Hopital Sud), Amiens
  - CHU Bordeaux, Bordeaux
  - CHU Cavale Blanche, Brest
  - Centre Fran ois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - H pital Beaujon, Clichy
  - Centre Georges-Fran ois Leclerc, Dijon
  - Grenoble University Hospital (Centre Hospitalier Universitaire Grenoble Alpes), La Tronche
  - CHU de LILLE - H pital HURIEZ, Lille
  - Hepatology, Hopital de la Croix-Rousse - 103 grande rue de la Croix-Rousse, Lyon
  - Centre L on B rard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie - Centre de Recherche, Paris
  - APHP Hospital Saint-Antoine, Paris
  - AP-HP Universit de Paris, Port Royal, Paris
  - Hopital Europeen Georges-Pompidou (HEGP), Paris
  - Hopital de la Croix Saint-Simon, Paris
  - Centre Hospitalier Universitaire de Bordeaux (CHU Bordeaux)(Hopitaux de Bordeaux) - Groupe hospitalier Sud - Hopital Haut-Levequ, Pessac
  - Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers
  - Insitute de Canc rologie de l'Ouest - Centre Ren Gauducheau, Saint-Herblain
  - ICANs, Strasbourg
  - Gustave Roussy Institute (IGR), Villejuif
- Italy (3):
  - Clinica Oncologica AOU (Azienda Ospedaliero Universitaria) delle Marche, Ancona
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Fondazione Policlinico Gemelli IRCCS, Rome
- Japan (15):
  - Eisai#1005, Nagoya, Aichi-ken
  - Eisai#1011, Toyoake, Aichi-ken
  - Eisai#1002, Kashiwa, Chiba
  - Eisai#1008, Matsuyama, Ehime
  - Eisai#1007, Kurume, Fukuoka
  - Eisai#1013, Akashi, Hyōgo
  - Eisai#1010, Kawasaki, Kanagawa
  - Eisai#1012, Kamigyō-ku, Kyoto
  - Eisai#1003, Sayama, Osaka
  - Eisai#1009, Hidaka, Saitama
  - Eisai#1001, Chuo-ku, Tokyo
  - Eisai#1006, Koto-ku, Tokyo
  - Eisai#1015, Minato-ku, Tokyo
  - Eisai#1004, Chiba
  - Eisai#1014, Niigata
- South Korea (9):
  - Korea University Guro Hospital, Guro-gu
  - National Cancer Center, Ilsandong-gu
  - Seoul National University Hospital, Jongno-gu
  - Seoul St. Mary's Hospital, Seocho-Gu
  - Severance Hospital (Yonsei University Medical Center), Seodaemun
  - Seoul National University Bundang Hospital, Seongnamsi Bundang
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Songpa-Gu
  - University of Ulsan College of Medicine - Asan Medical Center (AMC), Songpa-gu
- Spain (6):
  - University Hospital A Coru a, A Coruña
  - Fundaci Privada Institut d Investigaci Oncol gica de Vall-Hebron (VHIO), Barcelona
  - Hospital Universitario de Ja n, Jaén
  - Cl nica Universidad de Navarra, Madrid
  - H. Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (6):
  - Chang Gung Medical Foundation - Kaohsiung Branch, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Mesropian A, Gris-Oliver A, Balaseviciute U, Potdar AA, Kimura T, Shen J, Torres-Marcen M, Abril-Fornaguera J, Pique-Gili M, Camell-Raventos D, Peix J, Fernandez-Martinez E, Huguet-Pradell J, Hernandez de Sande A, Keraite I, Esteban-Fabro R, Barcena-Varela M, Lindblad KE, Lujambio A, Guccione E, Thung S, Ikeda M, Kudo M, Sia D, Pinyol R, Llovet JM. E7386 Enhances Lenvatinib's Antitumor Activity in Preclinical Models and Human Hepatocellular Carcinoma. Clin Cancer Res. 2025 Dec 1;31(23):5037-5050. doi: 10.1158/1078-0432.CCR-25-0725. PMID 40986544
- [Derived] Eskander RN, Lee JY, Mirza MR, Lorusso D, MacKay H, Ray-Coquard I, Oaknin A, Gonzalez-Martin A, Hasegawa K, Corr BR, Wu X, Leary A, Hu T, Dutta L, Okpara CE, McKenzie J, Makker V. Randomized study evaluating optimal dose, efficacy, and safety of E7386 plus lenvatinib versus treatment of physician's choice in advanced/recurrent endometrial carcinoma previously treated with platinum-based chemotherapy and immune checkpoint inhibitors. Int J Gynecol Cancer. 2025 Sep;35(9):101812. doi: 10.1016/j.ijgc.2025.101812. Epub 2025 Apr 5. PMID 40318924